CLINICAL TRIAL: NCT05210322
Title: The Percutaneous Cholangiopancreatoscopy Registry
Brief Title: Percutaneous Cholangiopancreatoscopy Registry
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00219877
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Biliary Stones; Cholangiocarcinoma, Intrahepatic; Biliary Stricture; Cholelithiasis; Choledocholithiasis
MeSH Terms: conditions — Cholecystolithiasis; Cholangiocarcinoma; Cholelithiasis; Choledocholithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Procedure: Percutaneous cholangiopancreatoscopy — Per standard treatment protocol for percutaneous cholangiopancreatoscopy, access will be gained into the biliary system using the biliary tube or into the gallbladder using the cholecystostomy tube. After access has been secured, through a peel-away sheath a Spy Glass Discover Digital Catheter will be introduced. Next, either, the stones will then be removed from the biliary system or gallbladder using a combination of baskets, and lithotripsy equipment as required, or in case of biliary strictures, a clamshell biopsy will be taken from the stricture site as identified on endoscopic visualization and cross-sectional imaging. Further intervention maybe performed for the stricture based on operator preference. After the complete stone removal/ stricture management the cholecystostomy/ biliary tube will be removed after the patient passes a clinical capping trial.

SUMMARY:
The Percutaneous Cholangiopancreatoscopy (PCPS) registry is an observational, multicentric, prospective, and retrospective registry of patients undergoing the percutaneous cholangiopancreatoscopy procedure at sites across the United States. In the retrospective component of the study, clinical and procedural data regarding patients who have undergone clinical indicated percutaneous cholangiopancreatoscopy procedure in the past will be collected from all the registry sites and stored in a secure database. The prospective component of the registry will run for three years at each site where patients undergoing the clinically indicated percutaneous cholangiopancreatoscopy procedure will be enrolled in the study, and the patients' data will be collected whenever the patients present to interventional radiology (IR) for a procedure or clinic visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults
* 18 years of age and older
* Patients undergoing clinically indicated percutaneous cholangiopancreatoscopy procedure at the Johns Hopkins Hospital or one of the registry sites.
* Willing and able to understand and sign a written informed consent document for the prospective component of the study.

Exclusion Criteria:

* Pregnant women
* Children (< 18 years of age)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with clinical indication for the cholangiopancreatoscopy procedure.
Sampling Method: Non-Probability Sample
Enrollment: 679 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Tube free survival | Up to 3 years
  Tube free survival will be calculated by estimating the number of patients who can undergo removal of the biliary/ cholecystostomy tube after the PCPS procedure until their last IR clinical follow-up or death.

SECONDARY OUTCOMES:
Technical success | At the time of the procedure
  Technical success is defined as successful access with cholangioscope and visualization of the stones or a lesion to be biopsied.
Procedural success | At the time of the procedure
  Procedural success in patients with calculi, is defined as either a) visualization of stones with at least partial stone removal, or b) visualization of biliary system demonstrating no need for further investigation; in patients with biliary stricture, defined as a) obtaining tissue for biopsy or b) successfully visualize and complete or partial treatment of the stricture.
Clinical success | At the time of the procedure
  Clinical success is defined as improvement in clinical symptoms (e.g., abdominal pain, fever, jaundice, nausea and vomiting), laboratory values and/or imaging findings.
Complication rate | At the time of the procedure
  Complication rate will be calculated by recording the adverse events that occur during the procedure in accordance with the Society of Interventional Radiology Classification System.
Complication rate | 1 month
  Complication rate will be calculated by recording the adverse events that occur after the procedure in accordance with the Society of Interventional Radiology Classification System.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Holly, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No